CLINICAL TRIAL: NCT03340155
Title: Explorative Investigations on the Mechanisms of Action of Photo(Chemo)Therapy in Skin Diseases
Brief Title: Mechanisms of Action of Photo(Chemo)Therapy in Skin Diseases
Acronym: BioUV2017
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Dermatology, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Graz IRB# 29-609 ex 16/17
Record Dates: First submitted 2017-10-29; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis; Cutaneous T Cell Lymphoma; Lymphoproliferative Disorders; Eczema; Lichen Planus; Prurigo; Pruritus; Polymorphic Light Eruption; Graft Vs Host Disease; Mastocytosis; Vitiligo
MeSH Terms: conditions — Psoriasis; Lymphoma, T-Cell, Cutaneous; Lymphoproliferative Disorders; Eczema; Lichen Planus; Prurigo; Pruritus; Graft vs Host Disease; Mastocytosis; Vitiligo

STUDY DESIGN:
Intervention Model Description: Biomarker search;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Photo(chemo)therapy — Treatment with photo(chemo)therapy, including UVB, UVA, PUVA and photopheresis

SUMMARY:
The molecular mechanisms of action of photo(chemo)therapy in skin diseases are investigated in this study. The phototherapeutic modalities employed include UVB (ultraviolet B), UVA (ultraviolet A), PUVA (psoralen+UVA) and/or extracorporeal photochemotherapy (photopheresis). The study will address whether and how photo(chemo)therapy affects specific biologic pathways in different skin disorders and search for predictive biomarkers.

DETAILED DESCRIPTION:
This study is performed in order to investigate the molecular mechanisms of action of photo(chemo)therapy in skin diseases, including psoriasis, cutaneous T-cell lymphoma, other lymphoproliferative disorders of the skin, eczema, lichen planus, prurigo/pruritus, polymorphic light eruption, mastocytosis, graft-versus-host disease, vitiligo and other photo(chemo)therapy-responsive diseases. Twenty patients will be enrolled per diagnosis group. The phototherapeutic modalities administered will be UVB, UVA, PUVA and/or extracorporeal photochemotherapy (photopheresis). The severity of disease and clinical response to treatment will be assessed with scores including dermatological quality of life (DLQI) and disease-specific scores such as PASI (psoriasis area and severity index), mSWAT (modified severity-weighted assessment tool), SCORAD (scoring atopic dermatitis), scleroderma score and/or different visual analog scale (VAS) scores for pruritus. The effect of treatment on a variety of laboratory endpoints will be investigated in blood samples and optionally also skin samples. Those endpoints include among others the regulation of cytokines/chemokines, immune function, clonality of immune cells, vitamin D, and serum lipids. The study will address whether and how photo(chemo)therapy affects specific biologic pathways in the different disorders and determine whether predictive biomarkers for therapeutic response exist.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Skin disorder to be treated with photo(chemo)therapy

Exclusion Criteria:

* Pregnancy and breastfeeding
* Poor general health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of soluble factors in the serum with clinical response, as measured by disease severity | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  Serum levels of cytokines, chemokine and other factors, as measured in pg/ml, will be correlated to the clinical response to treatment at the time points specified below to identify potential predictive biomarkers. Disease-specific scores such as PASI, mSWAT, SCORAD, scleroderma score and VAS pruritus scores will be used depending on the condition to carry-out correlation analysis, comparing the change from baseline to end of observation.
Correlation of cellular markers of peripheral lymphocytes with clinical response, as measured by disease severity | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  Expression of cellular markers including CD (cluster of differentiation) 1a, CD3, CD4, CD8, CD11c, CD25, CD45, CD56, CD68, CD103, CD163, FoxP3, as measured by flow cytometry will be correlated to the clinical response to treatment at the time points specified below to identify potential predictive biomarkers. Disease-specific scores such as PASI, mSWAT, SCORAD, scleroderma score and VAS pruritus scores will be used depending on the condition to carry-out correlation analysis, comparing the change from baseline to end of observation.
Evaluation of T cell receptor repertoire | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  Diversity of the T cell repertoire will be assessed by high-throughput sequencing of the T cell receptor and correlated to the clinical response to treatment at the time points specified below to identify its potential predictive value. Disease-specific scores such as PASI, mSWAT, SCORAD, scleroderma score and VAS pruritus scores will be used depending on the condition to carry-out correlation analysis, comparing the change from baseline to end of observation.

SECONDARY OUTCOMES:
Vitamin D concentration in serum | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  Vitamin D levels in serum will be assessed by immunoassay
Lipoprotein composition in serum | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  High density lipoprotein composition in serum will be investigated by proteomics and cholesterol efflux analysis
microRNA levels in serum | Day 14 to 0; week 4; week 8-12; week 12-16 (or month 6-12 for photopheresis)
  Levels of micro RNA (133, 206 207, 320, 99a, 150, 197 203 220, 423 and others) will be assessed by microarray assays

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Styria, Austria